CLINICAL TRIAL: NCT06868355
Title: APACE - Feasibility of Using Accelerometers to Measure Physical Activity in Cancer Patients on Early Phase Clinical Trials. A Feasibility Study Evaluating the Use of Accelerometers to Capture Physical Activity Levels in Cancer Patients on Early Phase Clinical Trials
Brief Title: APACE - Feasibility of Using Accelerometers to Measure Physical Activity in Cancer Patients on Early Phase Clinical Trials
Acronym: APACE
Status: Recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: The Christie NHS Foundation Trust (Other); Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Principal Investigator, Donna Graham, Medical Oncology Consultant, University of Manchester
Other Study IDs: NHS002002; 311863 (Other: IRAS)
Record Dates: First submitted 2025-02-25; First posted 2025-03-10 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Other: No intervention (observational study) — This is an observational study

SUMMARY:
Increased physical activity has been shown to improve outcomes for cancer patients, however the measure of activity is highly variable and understudied in cancer patients on early phase clinical trials where activity is used as a criteria for eligibility. Additionally, more than half of cancer patients experience fatigue at some point in their treatment with exercise and psychosocial interventions currently recommended as interventions. Therefore, it is important to be able to more accurately measure activity and fatigue in cancer patients to ensure adequate intervention, management and appropriate access to treatment.

This proposal is a non-interventional feasibility study designed to collect activity and sleep data from patients with advanced cancer newly enrolled in early phase clinical trials. The data will be collected over a 5-6 week period using a wearable accelerometer device. This study will be conducted concurrently with the early phase trial related activities/treatment and will have no impact on a patient's clinical pathway. Data generated from the study will be used to evaluate the feasibility of collecting activity and sleep data from patients with advanced cancer on early phase clinical trials.

In this study, participants in the UK will be able to opt-in to using eNutri, a web-based graphical food frequency questionnaire (FFQ), and provide feedback on its usability. The output of eNUTRI will help us understand if there is a use for eNutri in cancer care environments for a range of purposes such as providing nutritional support for cancer patients, and exploring drug-nutrient interactions on the patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary informed consent.
* Aged at least 16 years.
* Consented to an early phase clinical trial.
* Willingness to wear a device for the duration of the study.
* Willingness to comply with scheduled study procedures.
* ECOG PS 0 or 1.

Exclusion Criteria:

* Judgement by the investigator that the individual should not participate if they are unlikely to comply with study procedures and requirements.
* Patient deemed ineligible for enrolment onto an early phase clinical trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be identified by the research team for the Phase 1 study they are enrolling on; the Phase 1 study team are the participant's direct care team.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Minimum of 3 valid days of data per week or per study period. A valid day is defined as 16 hours of data across one day. | From baseline for a period of 4-8 weeks
  This data is collected by the accelerometer. A minimum of 3 valid days of data per week or study period indicates compliance of patients to protocol-defined use of accelerometers.
Successful return of both devices | From baseline for a period of 4-8 weeks
  Successful return of both devices indicates compliance of patients to protocol-defined use of accelerometers.

SECONDARY OUTCOMES:
Overall daily patient physical activity across 24 hours measured in millgravity | From baseline for a period of 4-8 weeks
  Accelerometer-collected activities will be summarised into the following statistic: Overall daily patient physical activity across 24 hour measured in milligravity. This statistic is a continuous variable and its agreement with patient-reported physical activity and investigator-assessed Eastern Cooperative Oncology Group Performance Status (ECOG PS) will be assessed using Pearson's correlation coefficient and one-way ANOVA.
Time spent in inactivity (total and in >30 minute periods over 24 hours) | From baseline for a period of 4-8 weeks
  This data is collected by the accelerometer. It is a continuous variable and its agreement with patient-reported physical activity and investigator assessed Eastern Cooperative Oncology Group Performance Status (ECOG PS) will be assessed using Pearson's correlation coefficient and one-way ANOVA.
Time spent in accelerometer-defined light intensity activity, moderate activity and vigorous activity throughout the day in minutes | From baseline for a period of 4-8 weeks
  This data is collected by the accelerometer. This statistic is a continuous variable and its agreement with patient-reported physical activity and investigator-assessed Eastern Cooperative Oncology Group Performance Status (ECOG PS) will be assessed using Pearson's correlation coefficient and one-way ANOVA.
Eastern Cooperative Oncology Group Performance Status (ECOG PS) as determined by investigator at each timepoint on the study | From baseline for a period of 4-8 weeks
  Patient-reported physical activity (captured from questionnaire) and investigator-assessed Eastern Cooperative Oncology Group Performance Status (ECOG PS) are categorical statistics. Their agreement will be assessed using Fisher's exact test.
Patient self-reported physical activity level (captured from questionnaire) | From baseline for a period of 4-8 weeks
  Patient-reported physical activity (captured from questionnaire) and investigator-assessed Eastern Cooperative Oncology Group Performance Status (ECOG PS) are categorical statistics. Their agreement will be assessed using Fisher's exact test.
The amount of time slept each night in minutes | From baseline for a period of 4-8 weeks
  This data is collected by the accelerometer. This statistic is a continuous variable and its agreement with patient's self-reported insomnia and investigator assessed insomnia will be assessed using Pearson's correlation coefficient and one-way ANOVA.
Sleep efficiency determined by calculating the time asleep (minutes) over the time spent in bed | From baseline for a period of 4-8 weeks
  This data is collected by the accelerometer. This statistic is a continuous variable and its agreement with patient's self-reported insomnia and investigator assessed insomnia will be assessed using Pearson's correlation coefficient and one-way ANOVA.
The variability in sleep duration over the study period | From baseline for a period of 4-8 weeks
  This data is collected by the accelerometer. This statistic is a continuous variable and its agreement with patient's self-reported insomnia and investigator assessed insomnia will be assessed using Pearson's correlation coefficient and one-way ANOVA.
Sleep regularity over the study period | From baseline for a period of 4-8 weeks
  This data is collected by the accelerometer. Sleep regularity over the study period is defined as the percentage probability of an individual being in the same state (asleep vs. awake) at any two time-points 24 hours apart. For example, if it is someone who works varying shift patterns sleep regularity would be low, e.g. they may be sleeping at midnight one day, but awake and working at that time the next day. Someone who goes to sleep and gets up at the same time each day would have high sleep regularity (closer to 100%).
Variability of sleep over the study period | From baseline for a period of 4-8 weeks
  This data is collected by the accelerometer. Variability of sleep over the study period is defined as follows: the sleep midpoint is the mid-point between sleep onset and waking. For each participant, we present the mean of this across all valid nights and the variability (standard deviation) across all valid nights. The standard deviation across all valid nights is the variability in sleep mid-point in minutes.
Documented insomnia grade by Common Terminology Criteria for Adverse Events (CTCAE) criteria | From baseline for a period of 4-8 weeks
  Investigator assessed insomnia grade by Common Terminology Criteria for Adverse Events (CTCAE) criteria and self-reported insomnia score (captured from questionnaire) are categorical statistics. Their agreement will be assessed using Fisher's exact test.
Patient reported insomnia score (captured from questionnaire) | From baseline for a period of 4-8 weeks
  Investigator assessed insomnia grade by Common Terminology Criteria for Adverse Events (CTCAE) criteria and self-reported insomnia score (captured from questionnaire) are categorical statistics. Their agreement will be assessed using Fisher's exact test.
Patient reported fatigue score (captured from questionnaire) | From baseline for a period of 4-8 weeks
  Investigator assessed fatigue grade by Common Terminology Criteria for Adverse Events (CTCAE) criteria and self-reported fatigue score (captured from questionnaire) are categorical statistics. Their agreement will be assessed using Fisher's exact test.
Documented fatigue grade by Common Terminology Criteria for Adverse Events (CTCAE) criteria at each study timepoint | From baseline for a period of 4-8 weeks
  Investigator assessed fatigue grade by Common Terminology Criteria for Adverse Events (CTCAE) criteria and self-reported fatigue score (captured from questionnaire) are categorical statistics. Their agreement will be assessed using Fisher's exact test.

CONTACTS AND LOCATIONS:
Locations (8):
- National Cancer Institute of Milan (INT), Milan, Italy
- Spain (5):
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - START Madrid CIOCC, Madrid
  - START Madrid Fundación Jiménez Díaz (FJD) Quiron Salud Hospital, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Instituto de Investigación Sanitaria (INCLIVA), Valencia
- United Kingdom (2):
  - University Hospitals of Leicester NHS Trust, Leicester
  - The Christie NHS Foundation Trust, Manchester